CLINICAL TRIAL: NCT05759715
Title: Iris Color and Day-Night Changes in the Sympathovagal Ratio
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Şahbender Koç, MD Cardıologist, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 1099/9.3.2016
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Iris Diseases
Keywords: LF/HF ratio, iris color, melanin
MeSH Terms: conditions — Iris Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 2-0 darkbown-green (2-0 bg): Those with distinctively dark brown in the central area, slightly green in the peripheral area,
  Interventions: Other: Iris Color Measurement , LF/HF Measurement
- 1-0 lightbrown-green (1-0 bg).: Those with slightly dark brown in the central area and green in the peripheral area,
  Interventions: Other: Iris Color Measurement , LF/HF Measurement
- dark brown (1-1 db): Eyes with the same color structure in the central iris and the peripheral iris.
  Interventions: Other: Iris Color Measurement , LF/HF Measurement
- light brown (1-1 lb): Eyes with the same color structure in the central iris and the peripheral iris.
  Interventions: Other: Iris Color Measurement , LF/HF Measurement
- dark brown (2-0 b): Those with distinctively dark brown in the central iris area compared to the periphery .
  Interventions: Other: Iris Color Measurement , LF/HF Measurement
- slightly dark brown (1-0 b): Those with slightly dark brown (1-0 b) in the central iris area compared to the periphery .
  Interventions: Other: Iris Color Measurement , LF/HF Measurement

INTERVENTIONS:
Other: Iris Color Measurement , LF/HF Measurement — Iris Color Measurement (Photos were taken of the iris with a digital camera ) LF/ HF Measurement (Using the three-channel standard ambulatory Holter recording system)

SUMMARY:
Iris melanocytes are innervated by parasympathetic and sympathetic nerve endings. Light affects autonomic nervous system activity via the retino-hypothalamic pathway. The hypothesis that the day-to-night variations in the sympatovagal ratio (LF/HF) may differ among individuals with different brown iris patterns was tested.

DETAILED DESCRIPTION:
A total of 621 healthy adults, aged between 16 and 50, with brown eyes and not diagnosed with a disease that might affect the autonomous nerve system were included in the study. A digital camera was used to acquire iris photos. Subjects were grouped into iris color groups (2-0 bg, 1-0 bg, 1-1 db, 1-1 lb, 2-0 b, and 1-0 b). Iris photos were analyzed with Picture Color Analyzer RBG software. The Central/Peripheral (R/RGB) ratio was used for objective distinction between the groups. Using 24-h Holter ECG monitoring, the change in the sympathovagal ratio from day (between 07:00 and 23:00 hrs) to night (between 23:00 and 07:00 hrs) was determined with the formula [(Day - Night) LF/HF)/Day LF/HF].

ELIGIBILITY:
Inclusion Criteria:

A total of 650 healthy individuals between the ages of 16 and 50 .

Exclusion Criteria:

Diseases that could affect the autonomic nervous system; Obesity Obstructive sleep apnea syndrome Hypertension Diabetes mellitus Atrial fibrillation Coronary disease Heart failure Goiter, etc.

Ages: 16 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 650 healthy individuals between the ages of 16 and 50 who applied for cardiac examination and had normal findings were recruited for the study.
Sampling Method: Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
LF/HF ratio | one week
  low frequency (LF, 0.04-0.15 Hz) and high frequency (HF, 0.16-0.4 Hz) measurements were taken from day and night changes in the heart rate by using the frequency-domain analysis method.